CLINICAL TRIAL: NCT06604611
Title: Efficacy and Safety of Colchicine in Patients with Heart Failure with Preserved Ejection Fraction and Inflammation
Brief Title: Colchicine in Patients with Heart Failure with Preserved Ejection Fraction and Inflammation
Acronym: CHIPS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dongying Zhang (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Dongying Zhang, Director, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHIPS
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure; Heart Failure with Preserved Ejection Fraction (HFPEF); Chronic Inflammation; Inflammation; Colchicine
Keywords: Heart Failure; Heart Failure with Preserved Ejection Fraction (HFpEF); Inflammation
MeSH Terms: conditions — Heart Failure; Inflammation | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly 1:1 allocate into either a colchicine-treated group or a blank control group, and patients included in different centers will be uniformly randomized by the main centre.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine Treatment Group (Experimental): This group is intended to include 100 patients, all of the patients will be given 5mg of once-daily the colchicine treatment on top of the SGLT2i treatment
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet Once Daily
- Control Group (No Intervention): The group is intended to include 100 patients, all of the patients will be given standard SGLT2i treatment

INTERVENTIONS:
Drug: Colchicine 0.5 MG Oral Tablet Once Daily — The intervention in this study is colchicine, patients randomized to the experimental group will be given oral colchicine 5mg once a day in 12 weeks.
  Arms: Colchicine Treatment Group

SUMMARY:
The main purpose of the CHIPS trial is to evaluate the efficacy and safety of colchicine in heart failure with preserved ejection fraction (HFpEF) patients with inflammation, including the effects of colchicine on circulating inflammatory markers, cardiac structure, cardiac function, clinical symptoms and exercise capacity in HFpEF patients.

DETAILED DESCRIPTION:
HFpEF is a disease with complex pathophysiological mechanisms, and inflammation has been found to be strongly associated with the onset and progression of HFpEF. Anti-inflammatory treatments begin to cut a striking figure in cardiovascular disease therapy. The LoDoCo2 trial showed a significant prognostic improvement of colchicine in patients with chronic coronary artery disease, and the latest COLICA trial, showed that 8 weeks of colchicine treatment significantly reduced levels of circulating inflammatory markers in patients with decompensated heart failure without serious adverse effects. However, at present, the efficacy and safety of colchicine for the treatment of HFpEF remains unclear. The CHIPS trial is a multi-center, randomized, open-label clinical trial. The aim of the study is to evaluate the efficacy and safety of colchicine in patients with heart failure with preserved ejection fraction and inflammation. The investigators proposed to assess changes in KCCQ scores, NT-proBNP levels, echocardiography and plasma inflammatory marker levels in HFpEF patients treated with or without colchicine to evaluate the efficacy of colchicine in HFpEF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction measured by echocardiography ≥ 50%
* Objective evidence of structural of functional abnormalities measured by echocardiography: 1)LVMI≥95 g/m2 in female and ≥115 g/m2 in male or 2)LAVI greater than 29ml/m2 in sinus rhythm or greater than 40ml/m2 in atrial fibrillation or 3)Average E/e' greater than 14 or 4)TR velocity greater than 2.8 m/s
* Patients with elevated NT-proBNP levels 24 hours after discontinuing intravenous diuretics: ≥300 pg/ml in patients with sinus heart rate; ≥600 pg/ml in patients with atrial fibrillation
* Both outpatient and admitted patients can be considered for enrollment. All patients must occurred worsening heart failure event within 30 days prior to randomization and a current NYHA cardiac function class II-IV
* Patients with CRP levels greater than 2mg/L
* Patient agrees to join and signs a written informed consent form

Exclusion Criteria:

* Received colchicine treatment within one month prior to randomization
* Acute coronary syndrome within 3 months prior to randomization, or history of pacemaker implantation, PCI, CABG within 3 months
* eGFR less than 25 mL/min/1.73 m2
* Liver function Child-Pugh class B or C
* Patient has a history of previous allergy to colchicine or dapagliflozin / empagliflozin
* Heart failure due to the following reasons: pericardial disease, pericardial effusion, myocarditis, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, and other rare cardiomyopathies such as Fabry disease
* Combined diagnosis of gastric ulcer, ulcerative colitis, Crohn disease and other digestive disorders or combined gastrointestinal tumors
* Plan to undergo cardiac surgery such as coronary revascularization, radiofrequency ablation of arrhythmias, valve replacement or other surgical procedures
* Pregnant or breastfeeding women
* The patient who is cognitively impaired and is unable to accurately complete the assessment and completion of the KCCQ scale with the assistance of a physician
* Autoimmune diseases such as systemic lupus erythematosus, long-term adrenocorticotropic hormone treatment for other diseases such as Schihan syndrome, or need to accept immunosuppressive drugs and monoclonal antibodies such as IL-1 and IL-6
* Patient with combined active solid tumor or hematological malignancy
* Patient comorbidity with other conditions that may be confused with HFpEF symptoms, such as acute exacerbation of COPD
* Admission with a well-defined infection (symptoms or pathogenetic evidence of infection, and leukocytes greater than 10*109/L)
* Previously diagnosed with HFrEF (initial assessment of LVEF less than 40%) or diagnosed with LVimpEF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in KCCQ-CS scores | Up to 12 weeks
  Patients were assessed for symptom improvement by Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CS)
Change in 6-MWD | Up to 12 weeks
  Improvement in patients exercise capacity assessed by 6-minuet walk distance
Change in serum CRP levels | Up to 12 weeks
  Change in serum C-reactive protein levels

SECONDARY OUTCOMES:
Change in serum NT-proBNP levels | Up to 12 weeks
  Change in serum N-terminal pro-B-type natriuretic peptide levels
Change in serum IL-1β levels | Up to 12 weeks
  Change in serum interleukin-1β levels
Change in serum IL-6 levels | Up to 12 weeks
  Change in serum interleukin-6 levels
Change in serum TNF-α levels | Up to 12 weeks
  Change in serum tumor necrosis factor-α levels
Change in cardiac structure | Up to 12 weeks
  Left ventricular mass index (LVMI) measured by echocardiography
Change in cardiac structure | Up to 12 weeks
  Left atrial volume index (LAVI) measured by echocardiography
Change in cardiac structure | Up to 12 weeks
  Left ventricular end-diastolic diameter (LVEDD) measured by echocardiography
Change in cardiac function | Up to 12 weeks
  Tricuspid annular plane systolic excursion (TAPSE) measured by echocardiography
Change in cardiac function | Up to 12 weeks
  Right ventricular ejection fraction (RVEF) measured by echocardiography
Change in cardiac function | Up to 12 weeks
  Peak mitral inflow velocity and peak diastolic mitral annulus velocity measured by echocardiography
Change in cardiac function | Up to 12 weeks
  Early diastolic mitral annular tissue velocity (e') measured by echocardiography
Worsening heart failure events | Up to 12 weeks
  Time to first worsening heart failure events, including hospitalization due to heart failure or intravenous diuretic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, MD. Ph.D., Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The next study will be conducted at the end of this study, so the data cannot be shared.

REFERENCES:
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Nidorf SM, Fiolet ATL, Mosterd A, Eikelboom JW, Schut A, Opstal TSJ, The SHK, Xu XF, Ireland MA, Lenderink T, Latchem D, Hoogslag P, Jerzewski A, Nierop P, Whelan A, Hendriks R, Swart H, Schaap J, Kuijper AFM, van Hessen MWJ, Saklani P, Tan I, Thompson AG, Morton A, Judkins C, Bax WA, Dirksen M, Alings M, Hankey GJ, Budgeon CA, Tijssen JGP, Cornel JH, Thompson PL; LoDoCo2 Trial Investigators. Colchicine in Patients with Chronic Coronary Disease. N Engl J Med. 2020 Nov 5;383(19):1838-1847. doi: 10.1056/NEJMoa2021372. Epub 2020 Aug 31. PMID 32865380
- [Background] Pascual-Figal D, Nunez J, Perez-Martinez MT, Gonzalez-Juanatey JR, Taibo-Urquia M, Llacer-Iborra P, Delgado J, Villar S, Mirabet S, Aimo A, Riquelme-Perez A, Anguita-Sanchez M, Martinez-Selles M, Noguera-Velasco JA, Ibanez B, Bayes-Genis A. Colchicine in acutely decompensated heart failure: the COLICA trial. Eur Heart J. 2024 Dec 1;45(45):4826-4836. doi: 10.1093/eurheartj/ehae538. PMID 39211951